CLINICAL TRIAL: NCT06738069
Title: Frequency of Chronic Kidney Disease Among Pregnant Women At Assuit University Hospitals
Brief Title: Chronic Kidney Disease in Pregnant Females
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Makram Ibrahim Ahmed, Doctor, Assiut University
Other Study IDs: CKD in pregnancy
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-09

CONDITIONS: CKD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pregnant female with CKD: Pregnant female Newly discovered as chronic kidney disease by our study.inclusion criteria including age 18 or above who accept to precipitate this study.. exclusion criteria including female actually known as CKD and female refusing to precipitate in our study... this female confirmed as CKD by positive Alb/Cr ratio in 2 occasions with 3 months duration in between
  Interventions: Other: Participants are not assigned an intervention as a part of the study
- Healthy pregnant female: Pregnant female without ckd and Alb /Cr ratio was negative
  Interventions: Other: Participants are not assigned an intervention as a part of the study

INTERVENTIONS:
Other: Participants are not assigned an intervention as a part of the study — Participants are not assigned an intervention as a part of the study

SUMMARY:
Screening of Chronic Kidney Disease among pregnant women for early detection

DETAILED DESCRIPTION:
Normal pregnancy associated with plasma volume expansion and hormonal changes lead to an increase in GFR of 40% to 65% in first and second trimester , with decrease in GFR of approximately 15% to 20% in the third trimester . Chronic Kidney Disease (CKD) is defined as abnormalities of kidney structure or function, present for a minimum of 3 months, with significant health implications .CKD classification is based on Cause, GFR category (G1-G5), and Albuminuria category (A1-A3), abbreviated as CGA . CKD during pregnancy is a major health concern ,affecting up to 3% of women of reproductive age in high-income countries, but estimated prevalence may be as much as 50% higher in low and middle-income countries (LMICs). Pregnant women with CKD at high risk of adverse maternal and fetal outcome , including hypertension development or worsening ,Preeclampsia, eclampsia , Anemia , platelets abnormalities , worsening kidney function ,need for cesarean section ,Pregnancy loss ,stillbirth ,Preterm labor ,Intrauterine growth restriction . CKD if detected and treated early in its course, ESRD is often preventable, especially for high risk individuals. CKD is often unrecognizable and asymptomatic until it is in its later stages, when the chances of preventing kidney failure are limited. Therefore, in order to administer targeted therapeutic interventions . early identification and stratification of those at highest risk of CKD are urgently needed. Screening programs using state of the art point-of-care testing equipment with blood and urine samples can test for CKD both quickly and accurately

ELIGIBILITY:
Inclusion Criteria:

* -all pregnant women at antenatal care who came to Outpatient clinic at the Women's Health Hospital and Nephrology Outpatient Clinic at Assiut University Hospitals
* At age of 18 yrs old or above . -Who accept to participate with this study

Exclusion Criteria:

* Pregnant women who are known CKD.
* Pregnant women refuse to participate with this study .
* Pregnant women with Acute Kidney Injury .

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study population will consist of pregnant women aged 18 years and older who present to Assiut University Hospitals for routine antenatal care or are admitted for delivery. We will include women from all trimesters of pregnancy who can provide informed consent. Exclusion criteria will encompass those with a diagnosis of acute kidney injury, a history of kidney transplantation, or chronic conditions that may confound CKD assessment unless specifically included in the study. We aim to recruit a total coverage for one year from October 2024 to September 2025. This study will provide valuable insights into the frequency of chronic kidney disease among pregnant women in this setting.
Sampling Method: Non-Probability Sample
Enrollment: 497 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of CKD among pregnant women attending antenatal care who came to outpatient clinic at the Women's Health Hospital and Nephrology Outpatient Clinic at Assiut University Hospitals | Through study completion, an average of 3 years

SECONDARY OUTCOMES:
Causes of CKD among pregnant women attending antenatal care who came to Outpatient clinic at the Women's Health Hospital and Nephrology Outpatient Clinic at assuit University Hospitals | Through study completion, an average of 3 years

REFERENCES:
- [Background] Farrell DR, Vassalotti JA. Screening, identifying, and treating chronic kidney disease: why, who, when, how, and what? BMC Nephrol. 2024 Jan 25;25(1):34. doi: 10.1186/s12882-024-03466-5. PMID 38273240
- [Background] Maule SP, Ashworth DC, Blakey H, Osafo C, Moturi M, Chappell LC, Bramham K, Milln J. CKD and Pregnancy Outcomes in Africa: A Narrative Review. Kidney Int Rep. 2020 May 26;5(8):1342-1349. doi: 10.1016/j.ekir.2020.05.016. eCollection 2020 Aug. PMID 32775838
- [Background] Kovesdy CP. Epidemiology of chronic kidney disease: an update 2022. Kidney Int Suppl (2011). 2022 Apr;12(1):7-11. doi: 10.1016/j.kisu.2021.11.003. Epub 2022 Mar 18. PMID 35529086
- [Background] Vinturache A, Khalil A, Glob. Libr. Women's me d., ISSN: 1756-2228; DOI 10.3843/GLOWM.411323